CLINICAL TRIAL: NCT05389631
Title: The International Trifecta and Epic Valve-in-Valve Registry: Detailed Insights Into Management Strategies and Outcomes
Brief Title: Trifecta and Epic ViV Detailed Insights Into Management Strategies and Outcomes
Status: Completed | Type: Observational
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-0249 / SH 10702
Record Dates: First submitted 2022-04-01; First posted 2022-05-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Aortic Valve Disease
Keywords: VinV TAVI; Trifecta valve; Epic valve
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trifecta VinV: VinV TAVI procedure in patients who have previously received a Trifecta valve
  Interventions: Other: no intervention
- Epic VinV: VinV TAVI procedure in patients who have previously received an Epic valve
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Non-randomized, open label, non-interventional, multicenter registry to describe risk factors, management strategies, and clinical outcomes in patients undergoing Valve in Valve (ViV) transcatheter aortic valve implantation (TAVI) in a previously implanted Trifecta or Epic valve using retrospective registry data from large volume centers

DETAILED DESCRIPTION:
Anonymized pre-, intra-, and postoperative data will be collected from patients undergoing VinV TAVI in a previously implanted Trifecta™ valve, Trifecta™ GT, Epic™ or Epic™ Supra valve from the largest volume implanters of the Trifecta and Epic valve in Europe until June 2020. The data will be analyzed in order to give a comprehensive description of clinical outcomes for Trifecta VinV procedures, to identify preoperative risk factors for coronary obstruction, 30-day and 1-year mortality, and other major complications, and to analyze the effects of patient characteristics and / or protective maneuvers in order to prevent coronary obstruction.

Differences of Trifecta and Epic failed patients will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a TAVI VinV procedure post-Trifecta or Epic implantation
* Patients who underwent planned or unplanned concomitant percutaneous coronary intervention (PCI) during the index hospital admission will be included, as will those undergoing emergent conventional cardiac surgery.

Exclusion Criteria:

* 1. TAVI VinV post-implantation of an aortic valve bioprosthesis other than the Trifecta or Epic valve
* 2. Patients undergoing combined, multiple transcatheter valve procedures in addition to TAVI VinV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing VinV TAVI procedures who have previously received a Trifecta or Epic valve in large volume implantation centers until June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
composite endpoint of 30-day all-cause mortality and/or unplanned coronary obstruction | 30 days
  coronary obstruction defined as (1) coronary obstruction resulting in myocardial infarction and/or cardiogenic shock, or (2) coronary obstruction requiring emergent coronary intervention with or without pre-TAVI coronary protection.

SECONDARY OUTCOMES:
all-cause mortality | 30-days
patients with unplanned coronary obstruction | 30-days
  coronary obstruction defined as (1) coronary obstruction resulting in myocardial infarction and/or cardiogenic shock, or (2) coronary obstruction requiring emergent coronary intervention with or without pre-TAVI coronary protection.
freedom from Major Adverse Cardiac Events defined as death, myocardial infarction or stroke | day of discharge from hospital after receiving VinV TAVI or 30 days, whichever is earlier
freedom from Major Adverse Cardiac Events defined as death, myocardial infarction or stroke | 1 year
freedom from Major Adverse Cardiac Events defined as death, myocardial infarction or stroke | up to 60 months
freedom from each individual Major Adverse Cardiac Event endpoint | day of discharge from hospital after receiving VinV TAVI or 30 days, whichever is earlier
freedom from each individual Major Adverse Cardiac Event endpoint | 1 year
freedom from each individual Major Adverse Cardiac Event endpoint | up to 60 months
freedom from other major Valve Academic Research Consortium 2 (VARC2) complications | day of discharge from hospital after receiving VinV TAVI or 30 days, whichever is earlier
freedom from other major VARC2 complications | 1 year
freedom from other major VARC2 complications | up to 60 months
post-VinV hemodynamic performance including transvalvular gradient, effective orifice area and paravalvular leak rate | day of discharge from hospital after receiving VinV TAVI or 30 days, whichever is earlier
post-VinV hemodynamic performance including transvalvular gradient, effective orifice area and paravalvular leak rate | 1 year
post-VinV hemodynamic performance including transvalvular gradient, effective orifice area and paravalvular leak rate | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borger, MD, PhD, Study Chair — Leipzig Heart Center
Locations (5):
- University Hospitals Leuven, Leuven, Belgium
- Germany (3):
  - Heart Center Dresden University Hospital, Dresden
  - University Hospital Jena, Jena
  - Heart Center Leipzig University Hospital, Leipzig
- Catharina Hospital Eindhoven, Eindhoven, Netherlands

REFERENCES:
- [Derived] Raschpichler M, Abdel-Wahab M, Curzen N, Wilbring M, Dubois C, Lam K, Faerber G, Nagel J, Thiele H, Borger MA. The International TrifectaTM and EpicTM Valve-in-Valve Registry: Insights Into Clinical & Hemodynamic Outcomes. Catheter Cardiovasc Interv. 2025 Jun;105(7):1711-1718. doi: 10.1002/ccd.31492. Epub 2025 Mar 27. PMID 40148747